CLINICAL TRIAL: NCT03042130
Title: Treatment With IV Iron in Hospitalized Patients With Severe Heart Failure But Without Iron Deficiency
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no recruitment
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-16-HO-512-CTIL
Record Dates: First submitted 2017-01-17; First posted 2017-02-03 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care; ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron Carboxymaltose (Experimental): standard of care + double dose of IV iron ferinject
  the medicine will be given twice within one week.
  Interventions: Other: Standard of care; Drug: Iron Carboxymaltose
- control (Other): standard of care
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — standard of care
Drug: Iron Carboxymaltose — Two IV doses
  Other Names: Ferinject
  Arms: Iron Carboxymaltose

SUMMARY:
Patients with congestive heart failure, grade 3-4, in addition to the standard care, will be randomized 1:1. The study group will receive 2 doses of IV iron (Iron carboxymaltose). The control group will receive standard of care alone. The study will test for the effects of the additional IV iron on the symptoms, clinical picture and quality of life of the treated patients.

DETAILED DESCRIPTION:
Patients with congestive heart failure, grade 3-4, in addition to the standard care, will be randomized 1:1. The study group will receive 2 doses of IV iron (Iron carboxymaltose). The control group will receive standard of care alone. The study will test for the effects of the additional IV iron on the symptoms, clinical picture and quality of life of the treated patients. The parameters that will be measured will include clinical, lab, echo, and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure grade 3-4
* Heart echo EF< 40% (ejection fraction)
* Hb > 10 mg/dL
* Iron> 50 mic/dL
* Iron/ transferrin rate > 20%

Exclusion Criteria:

* Infection
* Acute ischemia
* Patients that didn't receive the standard of care during 3 days before investigational product administration
* Hemochromatosis
* Known allergy to one of the products of the investigational product.
* Macrocytic anemia
* Iron excess
* Pregnant women
* Mentally disabled patients which can't give their concent properly.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Functioning improvement | 5 days after second administration
  NYHA assesment (New York Heart Association (NYHA) Functional Classification)
Quality of life improvement | 5 days after second administration
  KCCQ questionnaires
Functioning improvement | 1 month after second administration
  NYHA assesment (New York Heart Association (NYHA) Functional Classification)
Quality of life improvement | 1 month after second administration
  KCCQ (The Kansas City Cardiomyopathy Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Oster, Dr., Principal Investigator — Physician - Internal Medicine
Locations (1):
- Department of internal medicine A, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No